CLINICAL TRIAL: NCT05231161
Title: Diagnostic Performance of Exercise Stress Tests for the Detection of Epicardial and Microvascular Coronary Artery Disease
Acronym: UZ Clear
Status: Completed | Type: Observational
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: Centro Cardiologico Monzino (Other)
Responsible Party: Principal Investigator, Carlos Collet, Co-director Cardiovascular Center OLV Aalst, Onze Lieve Vrouw Hospital
Other Study IDs: CRI-100
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Index of Microvascular Resistance — The invasive diagnostic procedure will be performed in at least one coronary artery. The left anterior descending coronary artery will be the preferred target vessel; however, if technical factors precluded guidewire-based assessment of this artery (e.g., tortuous anatomy), then the left circumflex or right coronary artery can be selected. In the case of multiple measurements per patient, the lowest FFR or highest IMR will be used for analysis. A coronary wire with a pressure and temperature sensor (PressureWire X, Abbott Vascular, Santa Clara, CA, USA) will be advanced to the mid to distal segment of the coronary artery. Bolus thermodilution technique with three 3-cc saline injections in rest and hyperemia will be used.
  Other Names: Fractional Flow Reserve

SUMMARY:
Prospective, single-arm, multicenter study of patients with an intermediate pre-test probability of CAD and positive exercise stress tests referred for invasive angiography. Patients underwent an invasive diagnostic procedure (IDP) with measurement of fractional flow reserve (FFR) and index of microvascular resistance (IMR) in at least one coronary vessel. The objective was to determine the false discovery rate (FDR) of cardiac exercise stress tests with both FFR and IMR as references.

DETAILED DESCRIPTION:
The Redefining the Diagnostic Performance of Non-invasive Tests for the Detection of Coronary Artery Disease: UZ Clear is an investigator-initiated, single-arm, multicenter, prospective study of patients presenting with chest pain with an intermediate probability of CAD. The intermediate pre-test probability of CAD was defined based on the European Society of Cardiology Guidelines as a score between 15% and 85% based on age, sex, and the nature of symptoms. All patients had a positive exercise stress test and were referred for an invasive evaluation. Patients underwent a study protocol with an invasive diagnostic procedure (IDP) consisting of measurements of FFR and IMR in at least one coronary vessel. Exclusion criteria are acute coronary syndromes, known coronary artery disease, previous myocardial infarction, previous revascularization, and abnormal baseline electrocardiogram (ECG). All data were centrally collected and analyzed by the core laboratory.

The primary objective was to determine the false discovery rate of exercise stress tests using an interventional diagnostic procedure (IDP) with indexes of epicardial (FFR) and microvascular resistance (IMR) as clinical references. The secondary objective was to assess the impact of an IDP accounting for the presence of CMD on the accuracy of exercise stress tests.

ELIGIBILITY:
Inclusion Criteria:

- 1. Stable angina-like chest pain (typical or atypical) with intermediate (15-85%) pre-test probability of coronary artery disease using the ESC criteria.

2. Positive non-invasive exercise test, or inconclusive stress with additional positive imaging.

Exclusion Criteria:

1. Age <30 or >80-year old
2. Acute coronary syndromes.
3. Known coronary artery disease
4. Inability to perform exercise tests.
5. Previous myocardial infarction.
6. Previous CABG/PCI
7. Left ventricular dysfunction EF <35% or NYHA class III-IV
8. Uncontrolled or recurrent ventricular tachycardia
9. Atrial fibrillation
10. Severe renal dysfunction, defined as an eGFR <30 ml/min/1.73m2
11. Contra-indication to adenosine (e.g. asthma bronchial, severe COPD)
12. Active cancer
13. Recent stroke
14. Cardiomyopathy (dilated, hypertrophic, amyloidosis, arrhythmogenic right ventricular dysplasia)
15. Left Bundle Branch Block or baseline ST-segment depression >1mm.
16. Congenital heart disease
17. More than moderate valve disease

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stable patients suspected of having coronary artery disease based on the presence of stable angina-like chest pain
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The primary objective was to determine the false discovery rate of exercise stress tests using an interventional diagnostic procedure (IDP) with indexes of epicardial (FFR) and microvascular resistance (IMR) as clinical references. | Immediately post-procedural
  Diagnostic performance of exercise tests with false discovery rate

SECONDARY OUTCOMES:
to assess the impact of an IDP accounting for the presence of CMD on the accuracy of exercise stress tests. | Immediately post-procedural
  Comparison of false discovery rates using QCA, FFR and IMR as gold standards

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Aalst, Aalst, Oost Vlanderen, Belgium

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not foressen